CLINICAL TRIAL: NCT01112111
Title: Conventional Step-up, Step Down and a Novel Stimulation Regime in Controlled Ovarian Stimulation of Older Than 30 Years PCOS Patients Undergoing IVF- A Prospective Randomized Study.
Brief Title: A Novel Stimulation Protocol and the Conventional Low Dose Step-up and Step Down Regimens
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Genesis Center for Fertility & Human Pre-Implantation Genetics (Other)
Responsible Party: Savvas Koundouros, Genesis Centre for Fertility and Human Pre-implantation Genetics
Other Study IDs: PCOS; PCOS2; livfe67
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: PCOS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 75 PCOS Patients - step up regime: Group A will be comprised of 75 patients and these will receive a low dose step stimulation regime
  Interventions: Drug: mode of gonadotropin administration
- 75 PCOS patients -step down regime: Group B will be comprised of 75 patients who will receive a step down regime of stimulation
  Interventions: Drug: mode of gonadotropin administration
- 75 PCOS patients - sequential regime: Group C will be comprised of 75 patients who will be treated using a sequential stimulation regime
  Interventions: Drug: mode of gonadotropin administration

INTERVENTIONS:
Drug: mode of gonadotropin administration — Low dose step-up administration Step down administration sequential administration

SUMMARY:
This study is designed to compare the efficacy of a novel stimulation protocol with the conventional low dose step-up and step down regimens in older than 30 years PCOS patients undergoing in vitro fertilisation. The novel regime was proposed under the basis of the combined effectiveness of the two standard protocols to induce a uniform follicular growth and forms a continuation to the author's previously published results examining a similar approach in younger PCOS candidates. In total 225 patients have been recruited for this study. The stimulation protocol will be assigned under the basis of prospective randomization using sealed and numbered envelopes. All patients will be down regulated using a desensitisation agent administered on day 2 of spontaneous or induced withdrawal bleeding. The initial dosage in the low dose step-up regimen (group A) will be 150 IU/d of FSH for the first 6 days followed by an increase of 75 IU thereafter. In the step-down regimen (group B) patients will administer a starting dose of 300 IU/d of FSH for the first 3 days followed by a decrease to 225 IU/d for the next 3 days. This dosage will be further decreased to 150 IU/d or sustained at 225 IU (according to the initial response) until the day of the hCG injection. Group C, patients received 225 IU on day 1 followed by a decrease to 150 IU on day 2. On day 3 the dosage will be increased back to 225 IU. This alternation of injection dosage will be followed until day 6. According to the initial ovarian response the dosage will be sustained at 225 IU/d or 150 IU/d until the day of the hCG injection. The 10,000 IU hCG will be administered when at least two follicles had reached a mean diameter of 18 mm and the serum E2 levels were consistent with the ultrasound findings. Egg retrieval will be undertaken at 35 hours after the administration of the hCG injection. Oocytes recovered will be inseminated 4 hours post egg collection. Patients will receive 3 embryos on the third day of development. The luteal phase will be supported by progesterone suppositories starting on the day of the egg collection. A positive outcome will be detected by a serum β-hCG analysis 13 days after embryo replacement. The presence of a fetal heart pulse on ultrasound 3 weeks later confirmed a clinical pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Failure to ovulate after CC treatment

  * Over than 30 years of age No Previous IVF attempts
* Patent Fallopian Tubes
* Normo-spermic partners

Exclusion Criteria:

* Secondary Infertility
* Younger than 30 years
* Older than 36 years
* Other infertility cause

Ages: 30 Years to 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: PCOS is defined as the presence of polycystic ovaries, described as enlarged under US with more than 10 cysts (2 and 8 mm) in mean diameter and symptoms of oligomenorhrea/ amenorhea, high LH/FSH ratio, obesity, hyperandrogenism hirsuitism and acnes), and withdrawal bleeding after administration of progesterone. All women had either failed to ovulate after receiving a maximum daily dosage of 100-150 mg of clomiphene citrate for 5 days or failed to conceive after at least three ovulatory cycles using CC or gonadotropin treatment. Other inclusion criteria included: patients between 30 and 36 years old with patent fallopian tubes, no previous IVF attempts, and nortmo-spermic partners.
Sampling Method: Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Pregnancy Rate | The primary outcome measure will be assessed upon completion of the study estimated to September 2010

SECONDARY OUTCOMES:
Ovarian Response | The secondary outcome measure will be assessed upon completion of the controlled ovarian stimulation and the egg collection procedures. This parameter will be made known at least 5 weeks prior to the primary outcome mesure being availablle

CONTACTS AND LOCATIONS:
Locations (1):
- Genesis Centre for Fertility and Human Pre-implantation Genetics, Limassol, Limassol District, Cyprus